CLINICAL TRIAL: NCT02149121
Title: A Randomized, Controlled, Double-Blind, Parallel-Group, Phase 3 Study to Compare the Pharmacokinetics, Efficacy and Safety Between CT-P10, Rituxan and MabThera in Patients With Rheumatoid Arthritis
Brief Title: PK Similarity Prospective Phase 3 Study in Patients With Rheumatoid Arthritis
Acronym: rituximab
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-P10 3.2; 2013-004555-21 (EudraCT Number)
Record Dates: First submitted 2014-05-23; First posted 2014-05-29 (Estimated); Results first posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2017-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — CT-P10; Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CT-P10 (Experimental): rituximab, CT-P10(experimental drug), 1000mg by intravenous infusion. 2 infusions with a 2-week interval between the first and second infusion
  Interventions: Biological: CT-P10
- Rituxan (Active Comparator): US-licensed referece product, 1000mg by intravenous infusion. 2 infusions with a 2-week interval between the first and second infusions
  Interventions: Biological: CT-P10; Drug: Rituxan
- MabThera (Active Comparator): EU-approved reference product, 1000mg by intravenous infusion. 2 infusions with a 2-week interval between the first and second infusions
  Interventions: Biological: CT-P10; Drug: MabThera

INTERVENTIONS:
Biological: CT-P10 — 1000mg by intravenous infusion. 2 infusions with a 2-week interval between the first and second infusion
  Other Names: rituximab
Drug: Rituxan — US-licensed reference product, 1000mg by intravenous infusion. 2 infusions with a 2-week interval between the first and second infusion
  Other Names: rituximab
  Arms: Rituxan
Drug: MabThera — EU-approved reference product, 1000mg by intravenous infusion. 2 infusions with a 2-week interval between the first and second infusion
  Other Names: rituximab
  Arms: MabThera

SUMMARY:
This is a Phase 3 Study to Compare the Pharmacokinetics, Efficacy and Safety between CT-P10, Rituxan and MabThera in Patients with Rheumatoid Arthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is male or female between 18 and 75 years old, inclusive.
2. Patient has a diagnosis of RA according to the revised 1987 ACR classification criteria (Arnett et al 1988) for at least 6 months prior to randomization.
3. Patient has active disease as defined by the presence of 6 or more swollen joints (of 66 assessed) and 6 or more tender joints (of 68 assessed), and serum CRP ≥1.5 mg/dL (≥15 mg/L) or an ESR ≥28 mm/hour.
4. Patient has experienced an inadequate response to previous or current treatment with the anti-TNF agents infliximab
5. Patient has a proper discontinuation period after treatment with interleukin-1 receptor (IL-1R) antagonist, interleukin-6 receptor (IL-6R) antibody, or abatacept.

Exclusion Criteria:

1. Patient has taken more than 2 biologic agents.
2. Patient has previously been administered Rituximab or participated in a Rituximab biosimilar study.
3. Patient has allergies or hypersensitivity to murine, chimeric, human, or humanized proteins.
4. Patient has current or past history of chronic infection with hepatitis B, hepatitis C, or infection with human immunodeficiency virus (HIV)-1 or -2 or who has a positive result to the screening test for these infections.
5. Patient has an infection requiring oral antibiotics 2 weeks before randomization, parenteral injection of antibiotics 4 weeks before randomization, other serious infection 6 months before randomization, a history of recurrent herpes zoster or other chronic or recurrent infection 6 weeks before randomization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: DaeHyun Yoo, M.D., Ph.D, Principal Investigator — Hanyang University

REFERENCES:
- [Derived] Shim SC, Bozic-Majstorovic L, Berrocal Kasay A, El-Khouri EC, Irazoque-Palazuelos F, Cons Molina FF, Medina-Rodriguez FG, Miranda P, Shesternya P, Chavez-Corrales J, Wiland P, Jeka S, Garmish O, Hrycaj P, Fomina N, Park W, Suh CH, Lee SJ, Lee SY, Bae YJ, Yoo DH. Efficacy and safety of switching from rituximab to biosimilar CT-P10 in rheumatoid arthritis: 72-week data from a randomized Phase 3 trial. Rheumatology (Oxford). 2019 Dec 1;58(12):2193-2202. doi: 10.1093/rheumatology/kez152. PMID 31184752
- [Derived] Suh CH, Yoo DH, Berrocal Kasay A, Chalouhi El-Khouri E, Cons Molina FF, Shesternya P, Miranda P, Medina-Rodriguez FG, Wiland P, Jeka S, Chavez-Corrales J, Linde T, Hrycaj P, Abello-Banfi M, Hospodarskyy I, Jaworski J, Piotrowski M, Brzosko M, Krogulec M, Shevchuk S, Calvo A, Andersone D, Park W, Shim SC, Lee SJ, Lee SY. Long-Term Efficacy and Safety of Biosimilar CT-P10 Versus Innovator Rituximab in Rheumatoid Arthritis: 48-Week Results from a Randomized Phase III Trial. BioDrugs. 2019 Feb;33(1):79-91. doi: 10.1007/s40259-018-00331-4. PMID 30719632
- [Derived] Park W, Bozic-Majstorovic L, Milakovic D, Berrocal Kasay A, El-Khouri EC, Irazoque-Palazuelos F, Molina FFC, Shesternya P, Miranda P, Medina-Rodriguez FG, Wiland P, Jeka S, Chavez-Corrales J, Garmish O, Linde T, Rekalov D, Hrycaj P, Krause A, Fomina N, Piura O, Abello-Banfi M, Suh CH, Shim SC, Lee SJ, Lee SY, Kim SH, Yoo DH. Comparison of biosimilar CT-P10 and innovator rituximab in patients with rheumatoid arthritis: a randomized controlled Phase 3 trial. MAbs. 2018 Aug/Sep;10(6):934-943. doi: 10.1080/19420862.2018.1487912. Epub 2018 Jul 16. PMID 30010481
- See also: Related Info — http://www.celltrion.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from 76 study centers (including 1 GCP noncompliant study center) in Europe, Asia Pacific, and Latin America.
Pre-assignment Details: A total of 495 participants were screened for the study. Of theses, 111 participants were excluded from the study due to screening failure and 384 participants were enrolled in the study. Of these 384 participants, 12 participants from the significantly GCP noncompliant study center were excluded from all analysis populations.
Groups:
- CT-P10 (Main Study Period): This group received 1000mg rituximab (CT-P10; experimental drug) by intravenous (IV) infusion. Each participant received up to 3 treatment courses (2 treatment courses in the Main Study Period, and 1 additional treatment course in the Extension Study Period), if they met predefined eligibility criteria. Each course consisted of 2 infusions with a 2-week interval between the first and second infusions of a 24-week course. Throughout the study, Methotrexate (MTX) (7.5-25 mg/week orally or parenterally) and folic acid (≥ 5 mg/week) were coadministered.
- Rituxan (Main Study Period): This group received 1000mg rituximab (Rituxan; US-licensed reference product) by IV infusion. Each participant received up to 3 treatment courses (2 treatment courses in the Main Study Period, and 1 additional treatment course in the Extension Study Period), if they met predefined eligibility criteria. Each course consisted of 2 infusions with a 2-week interval between the first and second infusions of a 24-week course. Throughout the study, MTX (7.5-25 mg/week orally or parenterally) and folic acid (≥ 5 mg/week) were coadministered.
- MabThera (Main Study Period): This group received 1000mg rituximab (MabThera; EU-approved reference product) by IV infusion. Each participant received up to 3 treatment courses (2 treatment courses in the Main Study Period, and 1 additional treatment course in the Extension Study Period), if they met predefined eligibility criteria. Each course consisted of 2 infusions with a 2-week interval between the first and second infusions of a 24-week course. Throughout the study, MTX (7.5-25 mg/week orally or parenterally) and folic acid (≥ 5 mg/week) were coadministered.
- CT-P10/CT-P10 (Extension Study Period): For the Extension Study Period, participants, who were assigned to receive CT-P10 with their first infusion in the Main Study Period, were considered as CT-P10/CT-P10 group and maintained CT-P10 for the treatment course of the Extension Study Period at Extension Week 0. This group received 1000mg rituximab (CT-P10; experimental drug) by IV infusion with a 2-week interval between the first and second infusions of a 24-week course in the Extension Study Period followed by 1000mg rituximab (CT-P10; experimental drug) infusions in the Main Study Period. Throughout the study, MTX (7.5-25 mg/week orally or parenterally) and folic acid (≥ 5 mg/week) were coadministered.
- Rituxan/Rituxan (Extension Study Period): For the Extension Study Period, participants, who were assigned to receive Rituxan with their first infusion in the Main Study Period, were randomized in a 1:1 ratio to Rituxan/Rituxan group and Rituxan/CT-P10 group at Extension Week 0. This group is for participants who were assigned as Rituxan/Rituxan group and received 1000mg rituximab (Rituxan; US-licensed reference product) by IV infusion with a 2-week interval between the first and second infusions of a 24-week course in the Extension Study Period followed by 1000mg rituximab (Rituxan; US-licensed reference product) infusions in the Main Study Period. Throughout the study, MTX (7.5-25 mg/week orally or parenterally) and folic acid (≥ 5 mg/week) were coadministered.
- Rituxan/CT-P10 (Extension Study Period): For the Extension Study Period, participants, who were assigned to receive Rituxan with their first infusion in the Main Study Period, were randomized in a 1:1 ratio to Rituxan/Rituxan group and Rituxan/CT-P10 group at Extension Week 0. This group is for participants who were assigned as Rituxan/CT-P10 group and received 1000mg rituximab (CT-P10; experimental drug) by IV infusion with a 2-week interval between the first and second infusions of a 24-week course in the Extension Study Period followed by 1000mg rituximab (Rituxan; US-licensed reference product) infusions in the Main Study Period. Throughout the study, MTX (7.5-25 mg/week orally or parenterally) and folic acid (≥ 5 mg/week) were coadministered.
- MabThera/CT-P10 (Extension Study Period): For the Extension Study Period, participants, who were assigned to receive MabThera with their first infusion in the Main Study Period, were considered as MabThera/CT-P10 group and received CT-P10 for the treatment course of the Extension Study Period at Extension Week 0. This group received 1000mg rituximab (CT-P10; experimental drug) by IV infusion with a 2-week interval between the first and second infusions of a 24-week course in the Extension Study Period followed by 1000mg rituximab (Rituxan; US-licensed reference product) infusions in the Main Study Period. Throughout the study, MTX (7.5-25 mg/week orally or parenterally) and folic acid (≥ 5 mg/week) were coadministered.
Period: Main Study Period
Arm/Group | CT-P10 (Main Study Period) | Rituxan (Main Study Period) | MabThera (Main Study Period) | CT-P10/CT-P10 (Extension Study Period) | Rituxan/Rituxan (Extension Study Period) | Rituxan/CT-P10 (Extension Study Period) | MabThera/CT-P10 (Extension Study Period)
Started | 161 | 151 | 60 | 0 | 0 | 0 | 0
Completed | 140 | 134 | 56 | 0 | 0 | 0 | 0
Not Completed | 21 | 17 | 4 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 5 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 5 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Developed any malignancy | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Unmet predefined eligibility criteria | 2 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Disease progression | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Extension Study Period
Arm/Group | CT-P10 (Main Study Period) | Rituxan (Main Study Period) | MabThera (Main Study Period) | CT-P10/CT-P10 (Extension Study Period) | Rituxan/Rituxan (Extension Study Period) | Rituxan/CT-P10 (Extension Study Period) | MabThera/CT-P10 (Extension Study Period)
Started | 0 (This group is for the Main Study Period, not for the Extension Study Period.) | 0 (This group is for the Main Study Period, not for the Extension Study Period.) | 0 (This group is for the Main Study Period, not for the Extension Study Period.) | 122 (Some participants did not initiate the Extension Study Period (CT-P10: 19, Rituxan: 8, MabThera: 9). From 19 patients in CT-P10 who did not initiate the extension study period, one patient did not initiate the treatment course but had been included to extension period and was monitored up to week 48) | 64 (Some participants did not initiate the Extension Study Period (CT-P10: 19, Rituxan: 8, MabThera: 9)) | 62 (Some participants did not initiate the Extension Study Period (CT-P10: 19, Rituxan: 8, MabThera: 9)) | 47 (Some participants did not initiate the Extension Study Period (CT-P10: 19, Rituxan: 8, MabThera: 9))
Completed | 0 | 0 | 0 | 121 | 64 | 60 | 47
Not Completed | 0 | 0 | 0 | 1 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- CT-P10 (Main Study Period): This group received 1000mg rituximab (CT-P10; experimental drug) by IV infusion. Each participant received up to 3 treatment courses (2 treatment courses in the Main Study Period, and 1 additional treatment course in the Extension Study Period), if they met predefined eligibility criteria. Each course consisted of 2 infusions with a 2-week interval between the first and second infusions of a 24-week course. Throughout the study, MTX (7.5-25 mg/week orally or parenterally) and folic acid (≥ 5 mg/week) were coadministered.
- Total: Total of all reporting groups
Arm/Group | CT-P10 (Main Study Period) | Rituxan (Main Study Period) | MabThera (Main Study Period) | CT-P10/CT-P10 (Extension Study Period) | Rituxan/Rituxan (Extension Study Period) | Rituxan/CT-P10 (Extension Study Period) | MabThera/CT-P10 (Extension Study Period) | Total
Number analyzed (Participants) | 161 | 151 | 60 | 122 | 64 | 62 | 47 | 667
Age, Categorical [Count of Participants; unit: Participants] — Population: Study is divided in 2 period (Main Study Period and Extension Study Period) and baseline measures were separately entered. Therefore, a row population differs from the Overall.
  Participants
    number analyzed (Participants) | 161 | 151 | 60 | 0 | 0 | 0 | 0 | 372
    <=18 years | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Between 18 and 65 years | 142 | 127 | 56 | 0 | 0 | 0 | 0 | 325
    >=65 years | 18 | 24 | 4 | 0 | 0 | 0 | 0 | 46
Age, Categorical [Count of Participants; unit: Participants] — Population: Study is divided in 2 period (Main Study Period and Extension Study Period) and baseline measures were separately entered. Therefore, a row population differs from the Overall
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 122 | 64 | 62 | 47 | 295
    <=18 years | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
    Between 18 and 65 years | 0 | 0 | 0 | 105 | 57 | 52 | 44 | 258
    >=65 years | 0 | 0 | 0 | 16 | 7 | 10 | 3 | 36
Age, Continuous [Median (Full Range); unit: years] — Population: Study is divided in 2 period (Main Study Period and Extension Study Period) and baseline measures were separately entered. Therefore, a row population differs from the Overall
  years
    number analyzed (Participants) | 161 | 151 | 60 | 0 | 0 | 0 | 0 | 372
    (all) | 53.0 [18 to 74] | 53.0 [21 to 74] | 51.5 [20 to 74] |  |  |  |  | 53.0 [18 to 74]
Age, Continuous [Median (Full Range); unit: years] — Population: Study is divided in 2 period (Main Study Period and Extension Study Period) and baseline measures were separately entered. Therefore, a row population differs from the Overall
  years
    number analyzed (Participants) | 0 | 0 | 0 | 122 | 64 | 62 | 47 | 295
    (all) |  |  |  | 52.5 [18 to 74] | 52.5 [24 to 68] | 53.0 [28 to 72] | 50.0 [20 to 69] | 52.0 [18 to 74]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Study is divided in 2 period (Main Study Period and Extension Study Period) and baseline measures were separately entered. Therefore, a row population differs from the Overall
  Participants
    number analyzed (Participants) | 161 | 151 | 60 | 0 | 0 | 0 | 0 | 372
    Female | 138 | 130 | 50 |  |  |  |  | 318
    Male | 23 | 21 | 10 |  |  |  |  | 54
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Study is divided in 2 period (Main Study Period and Extension Study Period) and baseline measures were separately entered. Therefore, a row population differs from the Overall
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 122 | 64 | 62 | 47 | 295
    Female |  |  |  | 100 | 54 | 55 | 40 | 249
    Male |  |  |  | 22 | 10 | 7 | 7 | 46

OUTCOME MEASURES:

1. Primary Outcome: Analysis of Serum AUC0-last of Rituximab During the 1st Course of the Main Study Period (Over the First 24 Weeks) (ANCOVA)
Description: For evaluation of pharmacokinetics (PK), the primary endpoint was defined as the analysis of serum AUC0-last, AUC0-inf and Cmax of rituximab during the 1st course of the Main Study Period (over the first 24 weeks). During the 1st course of the Main Study Period, blood samples for PK analysis were collected every week from Week 0 to Week 4, every 4 weeks from Week 4 to Week 16, followed by Week 24.
  AUC0-last: Area under the concentration-time curve from time to the last measurable concentration over both doses of the 1st course
Time Frame: over the first 24 weeks
Population: PK population - The PK analysis set for the Main Study Period consisted of all patients who received 2 full doses (Week 0 and Week 2) of the study drug and provided at least 1 post-treatment PK concentration result during the 1st course in the Main Study Period.
Measure: Geometric Least Squares Mean (Standard Error); unit: h*μg/mL
Arm/Group | CT-P10 (Main Study Period) | Rituxan (Main Study Period) | MabThera (Main Study Period)
Number analyzed (Participants) | 62 | 60 | 59
h*μg/mL | 162414.81 (1.073) | 167309.07 (1.073) | 172450.97 (1.075)
Statistical Analysis 1: Comparison: CT-P10 (Main Study Period) vs Rituxan (Main Study Period); Primary PK analysis were analyzed using analysis of covariance (ANCOVA) model with treatment group as a fixed effect and gender, region, race, prior anti TNF alpha blocker status, and RF or anti-CCP status fitted as covariates; Test type: Equivalence — The equivalence of PK was to be concluded if the 90% CI for the ratio of geometric means in AUC0-last, AUC0-inf, and Cmax was entirely contained within the PK equivalence bounds of 80% and 125% for the following comparisons: CT-P10 versus Rituxan, CT-P10 versus MabThera, and Rituxan versus MabThera; Ratio of geometric least squares means = 97.07, 90% CI 2-sided [88.08 to 106.99] — Point estimates (geometric least squares means and ratios of geometric means) were calculated by back-transforming the least squares means
Statistical Analysis 2: Comparison: CT-P10 (Main Study Period) vs MabThera (Main Study Period); Primary PK analysis were analyzed using an ANCOVA model with treatment group as a fixed effect and gender, region, race, prior anti TNF alpha blocker status, and RF or anti-CCP status fitted as covariates; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least squares means = 94.18, 90% CI 2-sided [85.40 to 103.86] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Rituxan (Main Study Period) vs MabThera (Main Study Period); [analysis description as in outcome 1, analysis 2]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least squares means = 103.07, 90% CI 2-sided [93.32 to 113.85] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Analysis of Serum AUC0-inf of Rituximab During the 1st Course of the Main Study Period (Over the First 24 Weeks) (ANCOVA)
Description: For evaluation of PK, the primary endpoint was defined as the analysis of serum AUC0-last, AUC0-inf and Cmax of rituximab during the 1st course of the Main Study Period (over the first 24 weeks). During the 1st course of the Main Study Period, blood samples for PK analysis were collected every week from Week 0 to Week 4, every 4 weeks from Week 4 to Week 16, followed by Week 24.
  AUC0-inf: Area under the concentration-time curve from time 0 extrapolated to infinity over both doses of the 1st course
Time Frame: at Week 24 of the Main Study Period
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: h*μg/mL
Arm/Group | CT-P10 (Main Study Period) | Rituxan (Main Study Period) | MabThera (Main Study Period)
Number analyzed (Participants) | 59 | 60 | 56
h*μg/mL | 162377.28 (1.068) | 169480.80 (1.069) | 180637.81 (1.072)
Statistical Analysis 1: Comparison: CT-P10 (Main Study Period) vs Rituxan (Main Study Period); [analysis description as in outcome 1, analysis 2]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least squares means = 95.81, 90% CI 2-sided [87.39 to 105.04] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: CT-P10 (Main Study Period) vs MabThera (Main Study Period); [analysis description as in outcome 1, analysis 2]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least squares means = 89.89, 90% CI 2-sided [81.85 to 98.72] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Rituxan (Main Study Period) vs MabThera (Main Study Period); [analysis description as in outcome 1, analysis 2]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least squares means = 106.58, 90% CI 2-sided [97.03 to 117.08] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Analysis of Serum Cmax of Rituximab During the 1st Course of the Main Study Period (Over the First 24 Weeks) (ANCOVA)
Description: For evaluation of pharmacokinetics (PK), the primary endpoint was defined as the analysis of serum AUC0-last, AUC0-inf and Cmax of rituximab during the 1st course of the Main Study Period (over the first 24 weeks). During the 1st course of the Main Study Period, blood samples for PK analysis were collected every week from Week 0 to Week 4, every 4 weeks from Week 4 to Week 16, followed by Week 24.
  Cmax: Observed maximum concentration after the seocnd infusion of the 1st course
Time Frame: at Week 24 of the Main Study Period
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: ug/mL
Arm/Group | CT-P10 (Main Study Period) | Rituxan (Main Study Period) | MabThera (Main Study Period)
Number analyzed (Participants) | 62 | 59 | 59
ug/mL | 367.03 (1.042) | 386.65 (1.042) | 412.40 (1.043)
Statistical Analysis 1: Comparison: CT-P10 (Main Study Period) vs Rituxan (Main Study Period); [analysis description as in outcome 1, analysis 2]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least squares means = 94.92, 90% CI 2-sided [89.61 to 100.55] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: CT-P10 (Main Study Period) vs MabThera (Main Study Period); [analysis description as in outcome 1, analysis 2]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least squares means = 89.00, 90% CI 2-sided [84.01 to 94.28] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Rituxan (Main Study Period) vs MabThera (Main Study Period); [analysis description as in outcome 1, analysis 2]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least squares means = 106.66, 90% CI 2-sided [100.56 to 113.13] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Analysis of Change From Baseline of DAS28 (CRP) at Week 24 (ANCOVA)
Description: For evaluation of efficacy, the primary endpoint was defined as the analysis of change from baseline in disease activity measured by disease activity score 28 (DAS 28) C-reactive protein (CRP) at Week 24 between 2 treatment groups, CT-P10 and reference products (combined Rituxan and MabThera) groups. During the 1st course of the Main Study Period, DAS28 was assessed every 4 weeks from Week 0 to Week 24. DAS28 (CRP) was calculated using the following formula: DAS28 (CRP) = 0.56 X SQRT(TJC28) + 0.28 X SQRT(SJC28) + 0.36 X ln(CRP+1) + 0.014 X GH on VAS + 0.96. DAS28 (CRP) provides a number on a scale from 0 to 10 with higher values indicating greater RA disease activity.
Time Frame: at Week 24 of the Main Study Period
Population: Efficacy population - The efficacy analysis set for the Main Study Period consisted of all who received at least 1 full dose (1000mg) of study drug (CT-P10, Rituxan or MabThera), who had at least 1 post-treatment efficacy result and who did not have any major protocol violation including a violation of the inclusion and exclusion criteria.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Reference Products (Main Study Period): Reference products group: The combined Rituxan and MabThera groups. This group received 1000mg rituximab (Rituxan and MabThera) by IV infusion. Each participant received up to 3 treatment courses (2 treatment courses in the Main Study Period, and 1 additional treatment course in the Extension Study Period), if they met predefined eligibility criteria. Each course consisted of 2 infusions with a 2-week interval between the first and second infusions of a 24-week course. Throughout the study, MTX (7.5-25 mg/week orally or parenterally) and folic acid (≥ 5 mg/week) were coadministered.
Arm/Group | CT-P10 (Main Study Period) | Reference Products (Main Study Period)
Number analyzed (Participants) | 138 | 196
score on a scale | -2.11 (0.176) | -2.10 (0.178)
Statistical Analysis 1: Comparison: CT-P10 (Main Study Period) vs Reference Products (Main Study Period); Primary efficacy analysis were analyzed using an ANCOVA model with treatment group as a fixed effect and gender, region, race, study part, interaction of treatment group with study part, prior anti TNF alpha blocker status at baseline (intolerance case versus inadequate response), and RF or anti-CCP status fitted as covariates; Test type: Equivalence — Therapeutic equivalence was to be concluded if the 90% CI for the treatment difference in the change from baseline of DAS28 (CRP) at Week 24 was entirely within the equivalence margin of ±0.50; Mean Difference (Final Values) = -0.01, 90% CI 2-sided [-0.22 to 0.20] — Adjusted least squares means and standard error, estimate of treatment difference [CT-P10 - (Rituxan + MabThera)] and 2-sided 90% confidence interval calculated from the ANCOVA model

5. Secondary Outcome: Descriptive Statistics for Means (SD) for Baseline Value and Change From Baseline in Disease Activity Measured by DAS28 (CRP) of the Main Study Period
Description: For evaluation of efficacy, the secondary endpoint was defined as descriptive statistics of mean change from baseline in disease activity measured by DAS 28 (CRP) and DAS28 erythrocyte sedimentation rate (ESR) at Week 24 (efficacy population) and Week 48 (efficacy population - 2nd treatment course in Main Study Period subset) for the Main Study Period between 2 treatment groups, CT-P10 and reference products (combined Rituxan and MabThera) groups. DAS28 was assessed every 4 weeks from Week 0 to Week 24 during the 1st treatment course of the Main Study Period and every 8 weeks from Week 24 to Week 48 during the 2nd treatment course of the Main Study Period. DAS28 (CRP) was calculated using the following formula: DAS28 (CRP) = 0.56 X SQRT(TJC28) + 0.28 X SQRT(SJC28) + 0.36 X ln(CRP+1) + 0.014 X GH on VAS + 0.96. DAS28 (CRP) provides a number on a scale from 0 to 10 with higher values indicating greater RA disease activity.
Time Frame: at Week 24 of the Main Study Period
Population: Weeks 0 and 24 data were analysed by efficacy population who received at least 1 full dose of study drug and provided at least 1 post treatment efficacy result during 1st course. Week 48 data were analysed by 'efficacy-2nd course subset' who received at least 1 full dose and provided at least 1 post treatment efficacy result during 2nd course.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CT-P10 (Main Study Period) | Rituxan (Main Study Period) | MabThera (Main Study Period) | Reference Products (Main Study Period)
Number analyzed (Participants) | 155 | 144 | 59 | 203
score on a scale
  Week 0 (Baseline) | 5.8 (0.91) | 5.8 (0.92) | 6.0 (0.87) | 5.8 (0.91)
  Week 24 (1st course Week 24): number analyzed (Participants) | 138 | 138 | 58 | 196
  Week 24 (1st course Week 24) | -2.3 (1.06) | -2.3 (1.11) | -2.3 (1.30) | -2.3 (1.17)
  Week 48 (2nd course Week 24): number analyzed (Participants) | 131 | 128 | 54 | 182
  Week 48 (2nd course Week 24) | -2.7 (1.17) | -2.6 (1.32) | -2.7 (1.32) | -2.6 (1.32)

6. Secondary Outcome: Descriptive Statistics for Means (SD) for Baseline Value and Change From Baseline in Disease Activity Measured by DAS28 (CRP) of the Extension Study Period
Description: For evaluation of efficacy, the secondary endpoint was defined as descriptive statistics of mean change from baseline in disease activity measured by DAS28 (CRP) and DAS28 (ESR) at Week 72 (efficacy population-Extension Study Period subset) for the Extension Study Period between 4 treatment groups, CT-P10/CT-P10, Rituxan/Rituxan, Rituxan/CT-P10 and MabThera/CT-P10 groups. DAS28 was assessed every 8 weeks from Week 48 (Week 0 of the Extension Study Period) to Week 72 (Week 24 of the Extension Study Period) during the Extension Study Period. DAS28 (CRP) was calculated using the following formula: DAS28 (CRP) = 0.56 X SQRT(TJC28) + 0.28 X SQRT(SJC28) + 0.36 X ln(CRP+1) + 0.014 X GH on VAS + 0.96. DAS28 (CRP) provides a number on a scale from 0 to 10 with higher values indicating greater RA disease activity.
Time Frame: at Week 24 of the Main Study Period
Population: Efficacy - Extension Study Period subset: The "efficacy - Extension Study Period subset" consisted of all patients in the efficacy population who received at least 1 full dose (1000 mg) of study drug and provided at least 1 post-treatment efficacy result during the Extension Study Period.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Rituxan/Rituxan (Extension Study Period): For the Extension Study Period, participants, who were assigned to receive Rituxan with their first infusion in the Main Study Period, were randomized in a 1:1 ratio to Rituxan/Rituxan group and Rituxan/CT-P10 group at Extension Week 0. This group is for participants who were assigned as Rituxan/Rituxan group and received 1000mg rituximab (Rituxan; US licensed reference product) by IV infusion with a 2-week interval between the first and second infusions of a 24-week course in the Extension Study Period followed by 1000mg rituximab (Rituxan; US licensed reference product) infusions in the Main Study Period. Throughout the study, MTX (7.5-25 mg/week orally or parenterally) and folic acid (≥ 5 mg/week) were coadministered.
- Rituxan/CT-P10 (Extension Study Period): For the Extension Study Period, participants, who were assigned to receive Rituxan with their first infusion in the Main Study Period, were randomized in a 1:1 ratio to Rituxan/Rituxan group and Rituxan/CT-P10 group at Extension Week 0. This group is for participants who were assigned as Rituxan/CT-P10 group and received 1000mg rituximab (CT-P10; experimental drug) by IV infusion with a 2-week interval between the first and second infusions of a 24-week course in the Extension Study Period followed by 1000mg rituximab (Rituxan; US licensed reference product) infusions in the Main Study Period. Throughout the study, MTX (7.5-25 mg/week orally or parenterally) and folic acid (≥ 5 mg/week) were coadministered.
- MabThera/CT-P10 (Extension Study Period): For the Extension Study Period, participants, who were assigned to receive MabThera with their first infusion in the Main Study Period, were considered as MabThera/CT-P10 group and received CT-P10 for the treatment course of the Extension Study Period at Extension Week 0. This group received 1000mg rituximab (CT-P10; experimental drug) by IV infusion with a 2-week interval between the first and second infusions of a 24-week course in the Extension Study Period followed by 1000mg rituximab (Rituxan; US licensed reference product) infusions in the Main Study Period. Throughout the study, MTX (7.5-25 mg/week orally or parenterally) and folic acid (≥ 5 mg/week) were coadministered.
Arm/Group | CT-P10/CT-P10 (Extension Study Period) | Rituxan/Rituxan (Extension Study Period) | Rituxan/CT-P10 (Extension Study Period) | MabThera/CT-P10 (Extension Study Period)
Number analyzed (Participants) | 120 | 64 | 60 | 47
score on a scale | -3.0 (1.20) | -3.0 (1.32) | -2.9 (1.27) | -3.0 (1.11)

7. Secondary Outcome: Descriptive Statistics for Actual Value and Change From Baseline in Disease Activity Measured by DAS28 (ESR) of the Main Study Period
Description: For evaluation of efficacy, the secondary endpoint was defined as descriptive statistics of mean change from baseline in disease activity measured by DAS 28 (CRP) and DAS28 (ESR) at Week 24 (efficacy population) and Week 48 (efficacy population - 2nd treatment course in Main Study Period subset) for the Main Study Period between 2 treatment groups, CT-P10 and reference products (combined Rituxan and MabThera) groups. DAS28 was assessed every 4 weeks from Week 0 to Week 24 during the 1st treatment course of the Main Study Period and every 8 weeks from Week 24 to Week 48 during the 2nd treatment course of the Main Study Period. DAS28 (ESR) was calculated using the following formula: DAS28 (CRP) = 0.56 X SQRT(TJC28) + 0.28 X SQRT(SJC28) + 0.36 X ln(ESR) + 0.014 X GH on VAS. DAS28 (ESR) provides a number on a scale from 0 to 10 with higher values indicating greater RA disease activity.
Time Frame: at Week 24 of the Main Study Period
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Reference Products (Main Study Period): Reference products group: The combined Rituxan and MabThera groups. This group received 1000mg rituximab (Rituxan and MabThera) by IV infusion. Each participant received up to 3 treatment courses (2 treatment courses in the Main Study Period, and
  1 additional treatment course in the Extension Study Period), if they met predefined eligibility criteria. Each course consisted of 2 infusions with a 2-week interval between the first and second infusions of a 24-week course. Throughout the study, MTX(7.5-25 mg/week orally or parenterally) and folic acid (≥ 5 mg/week) were coadministered.
Arm/Group | CT-P10 (Main Study Period) | Rituxan (Main Study Period) | MabThera (Main Study Period) | Reference Products (Main Study Period)
Number analyzed (Participants) | 155 | 144 | 59 | 203
score on a scale
  Week 0 (Baseline) | 6.7 (0.83) | 6.7 (0.84) | 6.8 (0.75) | 6.7 (0.81)
  Week 24 (1st course Week 24): number analyzed (Participants) | 139 | 138 | 58 | 196
  Week 24 (1st course Week 24) | -2.5 (1.13) | -2.5 (1.13) | -2.3 (1.31) | -2.5 (1.18)
  Week 48 (2nd course Week 24): number analyzed (Participants) | 132 | 129 | 54 | 183
  Week 48 (2nd course Week 24) | -2.9 (1.29) | -2.8 (1.42) | -2.9 (1.32) | -2.8 (1.39)

8. Secondary Outcome: Descriptive Statistics for Actual Value and Change From Baseline in Disease Activity Measured by DAS28 (ESR) of the Extension Study Period
Description: For evaluation of efficacy, the secondary endpoint was defined as descriptive statistics of mean change from baseline in disease activity measured by DAS28 (CRP) and DAS28 (ESR) at Week 72 (efficacy population-Extension Study Period subset) for the Extension Study Period between 4 treatment groups, CT-P10/CT-P10, Rituxan/Rituxan, Rituxan/CT-P10 and MabThera/CT-P10 groups. DAS28 was assessed every 8 weeks from Week 48 (Week 0 of the Extension Study Period) to Week 72 (Week 24 of the Extension Study Period) during the Extension Study Period. DAS28 (ESR) was calculated using the following formula: DAS28 (CRP) = 0.56 X SQRT(TJC28) + 0.28 X SQRT(SJC28) + 0.36 X ln(ESR) + 0.014 X GH on VAS. DAS28 (ESR) provides a number on a scale from 0 to 10 with higher values indicating greater RA disease activity.
Time Frame: at Week 24 of the Main Study Period
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CT-P10/CT-P10 (Extension Study Period) | Rituxan/Rituxan (Extension Study Period) | Rituxan/CT-P10 (Extension Study Period) | MabThera/CT-P10 (Extension Study Period)
Number analyzed (Participants) | 120 | 64 | 60 | 47
score on a scale | -3.3 (1.24) | -3.3 (1.41) | -3.2 (1.36) | -3.2 (1.15)

9. Secondary Outcome: Analysis of B-cell Counts at Week 24 of the Main Study Period (ANCOVA)
Description: For evaluation of pharmacodynamics (PD), the endpoint was defined as B-cell counts at Week 24 between 2 treatment groups, CT-P10 and reference products (combined Rituxan and MabThera) groups. During the 1st course of the Main Study Period, B-cell kinetics blood samples were collected every week from Week 0 to Week 4, every 4 weeks from Week 4 to Week 16, followed by Week 24.
Time Frame: Week 24
Population: PD population - The PD analysis set for the Main Study Period consisted of all patients who received at least 1 full dose (1000mg) of study drug and provided at least 1 post-treatment PD result during the 1st course in the Main Study Period.
Measure: Geometric Least Squares Mean (Standard Error); unit: cells/mcL
Groups:
- CT-P10 (Main Study Period): This group received 1000mg rituximab (CT-P10; experimental drug) by IV) infusion. Each participant received up to 3 treatment courses (2 treatment courses in the Main Study Period, and 1 additional treatment course in the Extension Study Period), if they met predefined eligibility criteria. Each course consisted of 2 infusions with a 2-week interval between the first and second infusions of a 24-week course. Throughout the study, MTX (7.5-25 mg/week orally or parenterally) and folic acid (≥ 5 mg/week) were coadministered.
Arm/Group | CT-P10 (Main Study Period) | Reference Products (Main Study Period)
Number analyzed (Participants) | 123 | 173
cells/mcL | 25.29 (1.074) | 24.70 (1.073)
Statistical Analysis 1: Comparison: CT-P10 (Main Study Period) vs Reference Products (Main Study Period); Secondary PD analysis were analyzed using an ANCOVA model with results as the response, treatment group, as fixed effect and baseline values, gender, region, race, study part, interaction of treatment group with study part, prior anti-TNF alpha blocker status, and RF or anti-CCP status fitted as covariates; Test type: Other; Ratio of geometric least squares means = 102.37, 95% CI 2-sided [92.46 to 113.33]; Estimate of Geometric Least Square Mean and ratio of Geometric Least Square Means (CT-P10/reference products) were obtained from back transforming the least square means from the ANCOVA

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and adverse events (AEs) were assessed from the date the informed consent form was signed until the participant's last visit, up to week 24 of extension period (up to week 72).
Description: At each level of summarization, a participant is counted only once if they reported one or more events. Only the most severe event is counted. SAEs and AEs are considered to have occurred in the Main Study Period if start date is before the first infusion of the Extension Study Period or if participant did not enter the Extension Study Period, and considered to have occurred in the Extension Study Period if the start date is on or after the date of first infusion of the Extension Study Period.
Groups:
- CT-P10/CT-P10 (Extension Study Period): For the Extension Study Period, participants, who were assigned to receive CT-P10 with their first infusion in the Main Study Period, were considered as CT-P10/CT-P10 group and maintained CT-P10 for the treatment course of the Extension Study Period at Extension Week 0. This group received 1000mg rituximab (CT-P10; experimental drug) by IV infusion with a 2-week interval between the first and second infusions of a 24-week course. Throughout the study, MTX (7.5-25 mg/week orally or parenterally) and folic acid (≥ 5 mg/week) were coadministered.
- Rituxan/Rituxan (Extension Study Period): For the Extension Study Period, participants, who were assigned to receive Rituxan with their first infusion in the Main Study Period, were randomized in a 1:1 ratio to Rituxan/Rituxan group and Rituxan/CT-P10 group at Extension Week 0. This group received 1000mg rituximab (Rituxan; US-licensed reference product) by IV infusion with a 2-week interval between the first and second infusions of a 24-week course. Throughout the study, MTX (7.5-25 mg/week orally or parenterally) and folic acid (≥ 5 mg/week) were coadministered.
- Rituxan/CT-P10 (Extension Study Period): For the Extension Study Period, participants, who were assigned to receive Rituxan with their first infusion in the Main Study Period, were randomized in a 1:1 ratio to Rituxan/Rituxan group and Rituxan/CT-P10 group at Extension Week 0. This group received 1000mg rituximab (CT-P10) by IV infusion with a 2-week interval between the first and second infusions of a 24-week course. Throughout the study, MTX (7.5-25 mg/week orally or parenterally) and folic acid (≥ 5 mg/week) were coadministered.
- MabThera/CT-P10 (Extension Study Period): For the Extension Study Period, participants, who were assigned to receive MabThera with their first infusion in the Main Study Period, were considered as MabThera/CT-P10 group and received CT-P10 for the treatment course of the Extension Study Period at Extension Week 0. This group received 1000mg rituximab (CT-P10) by IV infusion with a 2-week interval between the first and second infusions of a 24-week course. Throughout the study, MTX (7.5-25 mg/week orally or parenterally) and folic acid (≥ 5 mg/week) were coadministered.
Arm/Group | CT-P10 (Main Study Period) | Rituxan (Main Study Period) | MabThera (Main Study Period) | CT-P10/CT-P10 (Extension Study Period) | Rituxan/Rituxan (Extension Study Period) | Rituxan/CT-P10 (Extension Study Period) | MabThera/CT-P10 (Extension Study Period)
All-Cause Mortality (participants affected / at risk) | 1/161 | 0/151 | 0/60 | 0/122 | 0/64 | 0/62 | 0/47
Serious Adverse Events (participants affected / at risk) | 13/161 | 14/151 | 4/60 | 4/122 | 0/64 | 1/62 | 0/47
Other Adverse Events (participants affected / at risk) | 88/161 | 72/151 | 29/60 | 27/122 | 16/64 | 17/62 | 7/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CT-P10 (Main Study Period) (N=161) | Rituxan (Main Study Period) (N=151) | MabThera (Main Study Period) (N=60) | CT-P10/CT-P10 (Extension Study Period) (N=122) | Rituxan/Rituxan (Extension Study Period) (N=64) | Rituxan/CT-P10 (Extension Study Period) (N=62) | MabThera/CT-P10 (Extension Study Period) (N=47)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — General disorders and administration site conditions
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CT-P10 (Main Study Period) (N=161) | Rituxan (Main Study Period) (N=151) | MabThera (Main Study Period) (N=60) | CT-P10/CT-P10 (Extension Study Period) (N=122) | Rituxan/Rituxan (Extension Study Period) (N=64) | Rituxan/CT-P10 (Extension Study Period) (N=62) | MabThera/CT-P10 (Extension Study Period) (N=47)
Upper respiratory tract infection (Infections and infestations) | 24 (32) | 30 (31) | 9 (12) | 10 (10) | 10 (10) | 8 (10) | 0 (0)
Urinary tract infection (Infections and infestations) | 15 (23) | 8 (14) | 2 (2) | 8 (10) | 2 (2) | 2 (3) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 10 (11) | 7 (9) | 3 (3) | 1 (1) | 3 (3) | 2 (2) | 2 (3)
Rhinitis (Infections and infestations) | 3 (4) | 6 (6) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infleunza (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion-related reaction (Injury, poisoning and procedural complications) | 33 (39) | 12 (15) | 13 (15) | 4 (5) | 3 (3) | 2 (2) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 5 (6) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (5) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 5 (5) | 7 (10) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 8 (9) | 8 (9) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 7 (7) | 4 (5) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 6 (7) | 5 (5) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 6 (6) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators could publish any information whatsoever and/or any discussion relating to Sponsor, Confidential Information, Inventions or work performed by investigator for Sponsor with the prior written consent of Sponsor.

DOCUMENTS (2):
  • Study Protocol (2016-04-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT02149121/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-02): https://cdn.clinicaltrials.gov/large-docs/21/NCT02149121/SAP_001.pdf